CLINICAL TRIAL: NCT03080506
Title: Effect of Elastic Abdominal Binder on Pain and Functional Recovery After Cesarean Delivery: a Randomized Controlled Trial
Brief Title: Abdominal Binder Following Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OBG-2559-04139
Record Dates: First submitted 2017-03-07; First posted 2017-03-15 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Cesarean Section Complications

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binder (Experimental): Each woman will be fitted with an elastic abdominal binder at the time of procedure completion just before leaving the operating room. The binder will be placed snuggly tight on top of the hospital gown at the infraumbilical level with the incision positioned at the middle part of the binder. The patients will be encouraged to wear binders at all time. However, periods of break from wearing the binder will be allowed at their convenience.
  Interventions: Device: Elastic abdominal binder
- No binder (No Intervention): The women will not be given a chance to wear abdominal binder or the likes.

INTERVENTIONS:
Device: Elastic abdominal binder — Participants will be fitted with an elastic abdominal binder at the time of procedure completion just before leaving the operating room. The binder will be placed snuggly tight on top of the hospital gown at the infraumbilical level with the incision positioned at the middle part of the binder. The patients will be encouraged to wear binders at all time. However, periods of break from wearing the binder will be allowed at their convenience.
  Arms: Binder

SUMMARY:
Cesarean delivery is a common obstetrical procedure and is associated with increased maternal morbidity and mortality. Pain and limited mobilization are major contributing factors that result in delayed functional recovery and complications. Elastic abdominal binder, a wide elastic belt that is wore around the patient's abdomen to support surgical incision after surgery, has been employed by clinicians for pain relief, wound complications prevention, improved pulmonary function, and stabilization. Benefits of the abdominal binder use have not been properly examined.

The aim of this study is to examine the effect of postcesarean elastic abdominal binder use on recovery by comparing pain scores and mobility function (through the 6-minute walk test [6MWT]) in postcesarean mothers who use versus do not use the elastic abdominal binder to support incisional site.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women undergoing cesarean delivery

Exclusion Criteria:

* Cesarean hysterectomy
* Intraoperative accidental injury to urinary or gastrointestinal organs
* Postoperative admission to intensive care unit (ICU)
* Postoperative intraperitoneal drain placement
* Unable to understand and follow oral/written instructions
* Severe neuromuscular or circulatory disorders
* Pulmonary diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2017-12-12 (Actual)

PRIMARY OUTCOMES:
Daily average postoperative pain scores | An average of pain scores at 8:00 am and 4:00 pm, up to 7 days postoperation
  A visual analog scale pain score
Postoperative functional recovery | In the morning of postoperative day 3
  Six-minute walk test (6MWT)

SECONDARY OUTCOMES:
Quality of life | In the morning of postoperative day 3
  The EuroQol Group's ED-5D-5L questionnaire
Postoperative complications | In the morning, up to 7 days postoperation
  Febrile morbidity, wound complications, bowel ileus

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, MSc, Study Chair — Chiang Mai University
Locations (1):
- Department of OB-GYN, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021